CLINICAL TRIAL: NCT04815941
Title: Effects of Soft Ball Tissue Release Exercises on Low Back Pain Secondary to Tight Hip Muscles.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/Lhr/1063
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Low Back Pain; Tight Hip Muscles
Keywords: Low Back Pain,Tight hip pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Soft ball tissue release exercises (Experimental)
  Interventions: Other: Soft ball tissue release exercises

INTERVENTIONS:
Other: Soft ball tissue release exercises — Exercise program were given to patients with low back pain secondary to hip muscle tightness using soft balls, i.e. tennis balls plus core stability exercises.
  3 days a week for four weeks.

SUMMARY:
It is also suggested that low back pain patients tend to have trigger point or tight muscles, i.e. Gluteus Maximus, Gluteus Medius, iliopsoas and Quardatus Lumborum, on at least one side.After approval from the university ethical committee, 23 (male, female) were enrolled in this study. All patients who presented nonspecific low back pain were included on the basis of inclusion and exclusion criteria. Demographic data of the patients were collected. Oswestry low back disability index was used to evaluate the disability level of low back. Piriformis muscle tightness was diagnosed among low back pain patients using FAIR (Flexion, abduction, internal rotation) and Freiberg's test. The FAIR test was performed on the patient in, side lying position, with the hip flexed at 60º and the knee flexed at 90º. With the hip being stabilized, a single examiner will internally rotate and adduct the hip by applying downward pressure onto the knee. Freiberg's test was performed on the patient in the supine position with the thigh extended. The leg and thigh are passively internally rotated by the examiner. If pain is registered, the test is positive. The effects of soft ball tissue release exercises on low back pain secondary to tight hip muscles

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-50 years Gender: Male and Female Low back pain for at least 12 weeks. Tight hip muscles (Priformis (FAIR test), TFL (Ober's test), Iliopsoas (Thomas test).

Exclusion Criteria:

* Any anatomical or neurophysiological causes of disease (X-ray and examination by a medical doctor) of spine.

Abnormal past histories of the spine, i.e. spondylitis, fracture, etc. Neurologic diseases. Functional restrictions on the upper and lower limbs. Disc prolapse Lumber Spinal stenosis L4-5 Spondylolysthesis Any abnormality at Sacroilliac joint (Faber,Pattricks,thigh thurst, ASIS distraction, Sacral compression test)

Ages: 35 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale | 2 months
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Neck disability Index | 2 months
  the overall score range is between 0 and 50, 0 being no to little pain and discomfort while 50 being the severest degree of pain and disability with complete activity limitation. The score is sometimes expressed in percentage as well.

CONTACTS AND LOCATIONS:
Overall Officials: Maryam Shabbir, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah Rehabilitation Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Geiger F, Bengtsson J, Berendse F, Weisser WW, Emmerson M, Morales MB, et al. Persistent negative effects of pesticides on biodiversity and biological control potential on European farmland. Basic and Applied Ecology. 2010;11(2):97-105.
- [Background] Casser HR, Seddigh S, Rauschmann M. Acute Lumbar Back Pain. Dtsch Arztebl Int. 2016 Apr 1;113(13):223-34. doi: 10.3238/arztebl.2016.0223. PMID 27120496
- [Background] Byrne DP, Mulhall KJ, Baker JF. Anatomy & biomechanics of the hip. The open sports medicine Journal. 2010;4(1).
- [Background] Heneweer H, Vanhees L, Picavet HS. Physical activity and low back pain: a U-shaped relation? Pain. 2009 May;143(1-2):21-5. doi: 10.1016/j.pain.2008.12.033. Epub 2009 Feb 12. PMID 19217208
- [Background] Boyajian-O'Neill LA, McClain RL, Coleman MK, Thomas PP. Diagnosis and management of piriformis syndrome: an osteopathic approach. J Am Osteopath Assoc. 2008 Nov;108(11):657-64. doi: 10.7556/jaoa.2008.108.11.657. PMID 19011229
- [Background] Hopayian K, Song F, Riera R, Sambandan S. The clinical features of the piriformis syndrome: a systematic review. Eur Spine J. 2010 Dec;19(12):2095-109. doi: 10.1007/s00586-010-1504-9. Epub 2010 Jul 3. PMID 20596735
- [Background] Durrani Z, Winnie AP. Piriformis muscle syndrome: an underdiagnosed cause of sciatica. J Pain Symptom Manage. 1991 Aug;6(6):374-9. doi: 10.1016/0885-3924(91)90029-4. PMID 1880438